CLINICAL TRIAL: NCT05060978
Title: Evaluation of the Effect of Two Online Interventions -Watch Your Weight During the Holidays Program and the Relative 5:2 Fasting- for the Prevention of Body Weight Gain at 8 Weeks in Mexican Adults in the Covid-19 Pandemic: A Pilot Three Arm Parallel-Group Randomized Controlled Trial
Brief Title: Evaluation of the Effect of Two Online Interventions -Watch Your Weight During the Holidays Program and the Relative 5:2 Fasting- for the Prevention of Body Weight Gain at 8 Weeks in Mexican Adults in the Covid-19 Pandemic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the retention of 78.1% of the participants obtained for the first measurement (after the December holidays), we believe that waiting one more year to complete the study would not be feasible for a subsequent definitive study.
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Research Professor, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USO313007128
Record Dates: First submitted 2021-09-27; First posted 2021-09-29 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Weight Gain; Overweight; Obesity
Keywords: Holiday Season; Normal weight; Prevention
MeSH Terms: conditions — Weight Gain; Overweight; Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Watch your Weight During the Holidays Program (Active Comparator)
  Interventions: Behavioral: Watch your Weight During the Holidays Program
- Relative 5:2 Fasting (Active Comparator)
  Interventions: Other: Relative 5:2 Fasting
- Control Group (Placebo Comparator)
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Watch your Weight During the Holidays Program — Participants in this group will have two video call individual sessions and one video call group session. This intervention will include self-monitoring strategies (self-weighing, diet monitoring and physical activity), and nutrition counseling and education. In addition, participants in this group will receive a weighing scale to achieve self-monitoring of body weight from the beginning of the study intervention until the end of the 52-weeks follow-up.
  Arms: Watch your Weight During the Holidays Program
Other: Relative 5:2 Fasting — Participants in this group will will have two video call individual sessions and one video call group session. This intervention will receive eating recommendations to follow a 5:2 intermittent fasting. They will be given low-calorie menus of 550 kcal and 660 kcal, for women and men respectively, which the participants in this group will apply on fasting days. The fasting will be held twice a week and on the remaining five days, the participants will not have any type of caloric restriction (it will be ad libitum). They will only have the general recommendation to adhere to a healthy dietary pattern.
  Arms: Relative 5:2 Fasting
Other: Control Group — Participants in this group will receive online information and a PDF file brochure during an individual video call session at the beginning of the 8-week period. This information will be about leading a healthy eating based on the norm for health promotion and education for healthy eating in Mexico (NOM-043-SSA2-2012).
  Arms: Control Group

SUMMARY:
Introduction. Obesity is the main risk factor for the development of chronic degenerative diseases in Mexico and other countries around the world. Due to the difficulty of treating obesity, it is necessary to change the curative paradigm for a preventive one. A review showed that holiday periods during the year are critical points for weight gain. The holiday season is the festive period with the greatest impact on adults' body weight. Observational studies have shown that more than 50% of the annual weight is gained during this period. However, few preventive interventions in the festive period have been carried out globally. Additionally, the COVID-19 pandemic seems to be negatively affecting diet, physical activity and body weight. So preventive interventions are needed, especially those that can be implemented in an online format. The purpose of the study is to evaluate the effect of two online interventions -Watch your Weight during the Holidays Program and the Relative 5:2 Fasting - on the prevention of body weight gain from baseline to 8 weeks in comparison with a control group in Mexican adults during the COVID-19 pandemic. Methodology: This is a Pilot Randomized Controlled Trial (RCT). The primary outcome is the change in body weight from baseline to 8 weeks. Secondary outcomes are the percentage of retention / desertion of the participants, adherence to interventions, participant satisfaction scale, changes in other obesity parameters, biochemical, physical, and quality of life variables from baseline to 8 weeks. Obesity and quality of life parameters from baseline to 52 weeks are also secondary outcomes. The statistical analysis of the primary and secondary variables will be conducted, according to their distribution, by intention to treat and, secondarily, by completer´s analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mexican adult participants (≥20 and ≤60 years)
* Residents of the city of Hermosillo, Sonora
* Body Mass Index ≥ 23 kg/m2 and ≤ 40 kg/m2
* Availability and motivation to attend the intervention program
* Committed to not undertake any other intervention in place of, or in combination with, the one assigned in the study during the 8 weeks of the intervention

Exclusion Criteria:

* Diagnosed medical conditions that constitute a contraindication for intervention such as: diabetes, hypertension, diseases with an effect on body weight (for example: liver failure; cancer in treatment or in advanced stage; history of COVID-19 that required hospitalization, supplemental oxygen or has left sequelae that contraindicates the intervention; psychiatric conditions; eating disorders, etc.).
* Use of drugs or substances with an effect on weight, for example, metformin, orlistat, corticosteroids, etc.
* Use of addictive substances such as drugs of abuse
* Previous bariatric surgery.
* Being a participant in another intervention or treatment for the management of obesity.
* Weight loss > 5% of total body weight in the last 4 months.
* Having plans to become pregnant within the study period, currently pregnant or breastfeeding.
* Another family member has agreed to participate in the study.
* Illiteracy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | Baseline to 8 weeks

SECONDARY OUTCOMES:
Changes in body weight | Baseline and 52 weeks
Changes in kilograms of body fat | Baseline, 8 weeks and 52 weeks
Changes in waist circumference | Baseline, 8 weeks and 52 weeks
Changes in systolic blood pressure | Baseline, 8 weeks and 52 weeks
Changes in diastolic blood pressure | Baseline, 8 weeks and 52 weeks
Changes in perception of health related quality of life | Baseline, 8 weeks and 52 weeks
  The SF-36 Health Survey evaluates aspects of the quality of life in adult populations (over 16 years of age). The result of its application is the generation of eight concepts or scales of health, result of the average of the sum of the questions contained in the questionnaire for each concept. These concepts are: physical function, physical role, corporal pain, general health, vitality, social function, emotional role and mental health. The SF-36 is a self-applied instrument and contains 36 questions. For each scale, the answers to each question are coded and recoded (10 questions), and the results are interpreted on a scale of 0 to 100, lower results indicate poorer health and greater result better health.
Retention / desertion | 8 weeks and 52 weeks
  The retention percentage will be obtained by dividing the number of people that finished the intervention the number that started the intervention, multiplied by 100. The dropout percentage will be obtained by the difference in the number of subjects who started and finished the intervention, multiplied by 100.
Adherence to intervention | 8 weeks and 52 weeks
  Adherence to the intervention will be calculated as the percentage of study measurement appointments and group sessions attended by each participant. Another way to measure adherence to interventions will be with a numerical scale of self-evaluation from 1 to 5, where 1 is the lowest score and 5 is the highest, to indicate how adherent they were to the meal plans.
Participant satisfaction scale | 8 weeks and 52 weeks
  Satisfaction of the participants in each of the intervention groups will be measured online using a scale from 1 to 5, where 1 is the lowest rating and 5 is the highest. A higher score means a higher satisfaction with the intervention recieved.
Changes in fasting glucose | Baseline and 8 weeks
Changes in total cholesterol | Baseline and 8 weeks
Changes in LDL cholesterol | Baseline and 8 weeks
Changes in HDL cholesterol | Baseline and 8 weeks
Changes in triglycerides | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rolando G Díaz Zavala, Ph.D., Principal Investigator — Universidad de Sonora
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora, Mexico